CLINICAL TRIAL: NCT06357247
Title: The Effect of SRS on Hemiplegia in Stroke Survivors: A Feasibility Study
Brief Title: The Effect of SRS on Hemiplegia in Stroke Survivors
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Feasibility and Funding, Planning to start enrolling again in early 2025
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: HM20027093
Record Dates: First submitted 2024-03-13; First posted 2024-04-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Stroke
Keywords: SRS- stochastic resonance stimulation; SR- stochastic resonance
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Feasibility Arm (Experimental): Wearing a stochastic resonance device at home in chronic stroke patients (six months or more post stroke).
  Interventions: Device: Sensory Threshold; Behavioral: Nine Hole Peg Test; Behavioral: Semmes Weinstein Monofilament Assessment

INTERVENTIONS:
Device: Sensory Threshold — Using a light, vibrotactile noise device on the participant's affected wrist. The actuator will be positioned on both the dorsal and volar sides of the wrist. Each participant's sensory threshold will be measured using the method of ascending and descending limits
Behavioral: Nine Hole Peg Test — The Nine-Hole Peg Test (NHPT) is considered as a gold standard measure of manual dexterity and most frequently used in MS research and clinical practice. The score for the 9-HPT is an average of the four trials. The two trials for each hand are averaged, converted to the reciprocals of the mean times for each hand and then the two reciprocals are averaged. On average, healthy male adults complete the NHPT in 19.0 seconds (SD 3.2) with the right hand, and in 20.6 seconds (SD 3.9) with the left hand.
Behavioral: Semmes Weinstein Monofilament Assessment — A non-invasive, low-cost, simple, and accurate handheld calibrated nylon thread that buckles once it has delivered a force of 10 g. It provides a standardized measure of a patient's ability to sense a point of pressure. The filaments are classified from grade 1 to 5 according to their thickness: 1.65-2.83 = grade 5, 3.22-3.61 = grade 4, 3.84-4.31 = grade 3, 4.56-6.45 = grade 2, and 6.65 = grade 1.

SUMMARY:
Strokes are one of the leading causes of long term disability and death in the United States. A stroke occurs when the blood supply to the brain is blocked, damaging parts of the brain. Many stroke survivors have difficulty completing dexterous hand movements and manipulating objects due brain damage in the sensorimotor cortex. Damage to these areas can cause decreased motor movements and tactile sensation on the affected side. Research shows that tactile sensation is necessary for maintaining grip, grading grip forces and decreasing object slippage. Therefore, it is important to address tactile sensation with motor performance during stroke rehabilitation to improve performance outcomes among stroke survivors.

DETAILED DESCRIPTION:
A novel intervention that has shown immediate improvements in tactile sensation is called stochastic resonance stimulation. SRS is a phenomenon where cutaneous sensation can be enhanced with the presence of tactile noise in a nonlinear system. This theory suggests that the application of an imperceptible vibrotactile stimulation increases the synchronization of afferent neurons firing to the somatosensory cortex, ultimately increasing the excitability of mechanoreceptors in the skin suggesting that afferent signals from the periphery to the somatosensory cortex influence motor movements. However, more research is needed to document the changes in motor performance with the use of SRS and it is unclear how SRS stimulation changes different measurable sensory processing differences

ELIGIBILITY:
Inclusion Criteria:

* Stroke survivors over the age of 18
* At least six months post stroke
* Ability to provide verbal informed consent and written informed consent
* Score of at least 56 on the Fugl meyer assessment total motor scores
* Able to detect at least 6.65 (300 grams) on the Semmes Weinstein monofilament on both the pads of the thumb and index finger
* Able to complete the nine hole peg test
* Able to reliably express pain, discomfort, or fear
* Speak english

Exclusion Criteria:

* History of upper extremity orthopedic conditions, such as arthritis, surgery, etc.
* Aphasia caused by stroke
* Does not have AROM
* Currently have muscle contractures in upper extremity
* Participating in other research studies
* Patients with electrically operated implanted device (e.g. cardiac pacemaker/defibrillator, drug delivery pump, and neurostimulator)
* History of SMI (e.g. schizophrenia, schizoaffective disorder)
* History of neurodegenerative disability (e.g. Multiple Sclerosis, Parkinson's Disease)
* Have received botulinum injections in the paretic limb within the past three months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-03-04 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Scores on ease of use, duration of wear, and preference related to wearing a stochastic resonance device at home in chronic stroke patients | Six months post stroke
  To determine the feasibility of wearing a stochastic resonance device at home in chronic stroke patients. This is administered through a participant questionnaire. Some questions are point-based (scale of 1-5), and some are open-ended questions. A good score is considered to be a higher signal-to-noise ratio, indicating better performance and detection capabilities

SECONDARY OUTCOMES:
Optimal level of stochastic resonance vibration | Six months post stroke
  To determine the optimal level of stochastic resonance vibration (120% vs 90% vs 60% of detection threshold) in stroke survivors

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Chu, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States